CLINICAL TRIAL: NCT05262660
Title: The Long-term Effect of Superselective Adrenal Arterial Embolization and Medical Treatment for Primary Aldosteronism on Cardiorenovascular Protection, Blood Pressure, and the Endocrinological Profile.
Brief Title: The Long-term Effect of SAAE and Medical Treatment for Primary Aldosteronism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: SAAE-001
Record Dates: First submitted 2022-01-09; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Primary Aldosteronism
Keywords: Adrenal Arterial Embolization; mineralocorticoid receptor antagonist; clinical outcomes
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — In-hospital data were obtained from the electronic medical record system (EMRS) at our institution. The 1-month ,6-month,12-month, 2-year and 3-year data were obtained from out-patient follow-up records in the EMRS, which included their complaints, antihypertensive regimens, office, and 24-hr mean blood pressures, biochemical parameters (plasma renin, aldosterone, and potassium), adverse events, and adrenal computerized tomography (only at 6 months). Clinical and biochemical outcomes were assessed based on Primary Aldosteronism Surgical Outcome (PASO) criteria and were classified as complete success, partial success, or absent success.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SAAE group: Patients who were diagnosed with primary aldosteronism choice SAAE at our institution
- MRA group: Patients who were diagnosed with primary aldosteronism choice medical treatment(mineralocorticoid receptor antagonists, MRA)) at our institution

SUMMARY:
In this prospective controlled trial, we aim to determine whether superselective adrenal artery embolization is superior to medical treatment for patients with PA who refuse surgery for medication. Patients age 18 to 75 years with hypertension will be screened for the presence of PA according to Endocrine Society Clinical Practice Guidelines. Patients with confirmed PA are counseled on the treatment option, including adrenalectomy. Those who opt to enroll in the study choice either SAAE or spironolactone (20-60mg daily) therapy (medical group). In both groups, if office blood pressure exceeds 140/90mmHg, amlodipine and terazosin will sequentially be added to the initial therapy form month 1 to year 3. The primary endpoint is the change in blood pressure, and the secondary end point is the change in biochemical outcomes. The Primary Aldosteronism Surgical Outcome criteria are used to classify clinical and biochemical outcomes as complete, partial, or absent success.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is the main cause of secondary hypertension, affecting 5%-15% of the general hypertensive population. Early diagnosis and treatment are of crucial importance because patients with PA are more susceptible to cardiovascular morbidity and mortality than primary hypertensive patients. Traditional treatments such as medication with mineralocorticoid receptor antagonists and adrenalectomy have some limitations. Over the past decade, superselective adrenal artery embolization (SAAE) has been used to treat PA, but their efficacies have not been compared with medication-controlled studies. Recent study found that SAAE is an effective and safe treatment for patients with PA. In this prospective controlled trial, we aim to determine whether this procedure is superior to medical treatment for patients with PA who refuse surgery for medication.

Patients age 18 to 75 years with hypertension will be screened for the presence of PA according to Endocrine Society Clinical Practice Guidelines. Adrenal computed tomography will be performed in all patients. Patients willing to participate in the study also will undergo adrenal venous sampling (AVS) Serum aldosterone and renin levels are measured by chemiluminescence immunoassay. Patients with confirmed PA are counseled on the treatment option, including adrenalectomy. Those who opt to enroll in the study choice either SAAE or spironolactone (20-60mg daily) therapy (medical group). In both groups, if office blood pressure exceeds 140/90mmHg, amlodipine and terazosin will sequentially be added to the initial therapy form month 1 to year 3. The primary endpoint is the change in blood pressure, and the secondary end point is the change in biochemical outcomes. The Primary Aldosteronism Surgical Outcome Criteria are used to classify clinical and biochemical outcomes as complete, partial, or absent success.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PA
* They refused medication treatment due to intolerance of side effects
* They had lateralization by adrenal venous sampling (AVS), and refused the adrenalectomy

Exclusion Criteria:

* History of serious contrast agent allergy
* Complication with severe liver diseases
* History of myocardial infarction and stent implantation within the past 3 months
* Renal insufficiency, with serum creatinine >176 umo/L
* Pregnancy or lactation
* History of participation in another clinical trial in the past 3 months
* Any serious comorbidity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients were willing to participate and then hospitalized for further evaluation. Antihypertensive medications that affect the renin-angiotensin-aldosterone system were stopped for two weeks, diuretics and MRA were withdrawn for at least 4 weeks before ARR testing. Hypertensive patients were prescribed with verapamil and/or terazosin based on Endocrine Society Clinical Practice Guideline. Patients with positive aldosterone-to-renin ratio underwent one of the following confirmatory tests: saline infusion test or captopril inhibition test. Adrenal CT scan and adrenal venous sampling (AVS) were performed for subtype classification of the PA. The PA patients were counseled on the various treatment options, including surgery, medications, and adrenal artery ablation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes-Change from Baseline Systolic Blood Pressure | at 12 months
  Complete clinical success is defined as normotension without the aid of antihypertensive medication. Partial clinical success is defined as the same blood pressure as before treatment with less antihypertensive medication or a reduction in blood pressure with either the same amount or less antihypertensive medication. Absent clinical success is defined as unchanged or increased blood pressure with either the same amount or an increase in antihypertensive medication
Clinical outcomes-Change from Baseline Systolic Blood Pressure | at 24 months
  Complete clinical success is defined as normotension without the aid of antihypertensive medication. Partial clinical success is defined as the same blood pressure as before treatment with less antihypertensive medication or a reduction in blood pressure with either the same amount or less antihypertensive medication. Absent clinical success is defined as unchanged or increased blood pressure with either the same amount or an increase in antihypertensive medication
Clinical outcomes-Change from Baseline Systolic Blood Pressure | at 36 months
  Complete clinical success is defined as normotension without the aid of antihypertensive medication. Partial clinical success is defined as the same blood pressure as before treatment with less antihypertensive medication or a reduction in blood pressure with either the same amount or less antihypertensive medication. Absent clinical success is defined as unchanged or increased blood pressure with either the same amount or an increase in antihypertensive medication

SECONDARY OUTCOMES:
biochemical outcomes-Change from Baseline hypokalaemia and the aldosterone/plasma renin | at 12 months
  Complete biochemical success is defined as correction of hypokalaemia (if present pretreatment) and normalization of the aldosterone/plasma renin(ARR); in patients with a raised ARR after treatment, aldosterone secretion should be suppressed in a confirmatory test. Partial biochemical success is defined as correction of hypokalaemia (if present pre-treatment) and a raised ARR with one or both of the following (compared with pre-treatment): ≥50% decrease in baseline plasma aldosterone concentration; or abnormal but improved post-treatment confirmatory test result. Absent biochemical success is defined as persistent hypokalaemia (if present pre-treatment) or persistent raised ARR, or both, with failure to suppress aldosterone secretion with a post-treatment confirmatory test
biochemical outcomes-Change from Baseline hypokalaemia and the aldosterone/plasma renin | at 24 months
  Complete biochemical success is defined as correction of hypokalaemia (if present pretreatment) and normalization of the aldosterone/plasma renin(ARR); in patients with a raised ARR after treatment, aldosterone secretion should be suppressed in a confirmatory test. Partial biochemical success is defined as correction of hypokalaemia (if present pre-treatment) and a raised ARR with one or both of the following (compared with pre-treatment): ≥50% decrease in baseline plasma aldosterone concentration; or abnormal but improved post-treatment confirmatory test result. Absent biochemical success is defined as persistent hypokalaemia (if present pre-treatment) or persistent raised ARR, or both, with failure to suppress aldosterone secretion with a post-treatment confirmatory test
biochemical outcomes-Change from Baseline hypokalaemia and the aldosterone/plasma renin | at 36 months
  Complete biochemical success is defined as correction of hypokalaemia (if present pretreatment) and normalization of the aldosterone/plasma renin(ARR); in patients with a raised ARR after treatment, aldosterone secretion should be suppressed in a confirmatory test. Partial biochemical success is defined as correction of hypokalaemia (if present pre-treatment) and a raised ARR with one or both of the following (compared with pre-treatment): ≥50% decrease in baseline plasma aldosterone concentration; or abnormal but improved post-treatment confirmatory test result. Absent biochemical success is defined as persistent hypokalaemia (if present pre-treatment) or persistent raised ARR, or both, with failure to suppress aldosterone secretion with a post-treatment confirmatory test

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiu Yang, Study Chair — First Affiliated Hospital of Chengdu Medical College
Locations (1):
- Yaqiong Zhou, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang H, Li Q, Liu X, Zhao Z, He H, Sun F, Hong Y, Zhou X, Li Y, Shen R, Bu X, Yan Z, Zheng H, Yang G, Zhu Z; Chongqing Endocrine Hypertension Collaborative Team. Adrenal artery ablation for primary aldosteronism without apparent aldosteronoma: An efficacy and safety, proof-of-principle trial. J Clin Hypertens (Greenwich). 2020 Sep;22(9):1618-1626. doi: 10.1111/jch.13960. Epub 2020 Aug 27. PMID 32852871
- [Result] Zhao Z, Liu X, Zhang H, Li Q, He H, Yan Z, Sun F, Li Y, Zhou X, Bu X, Wu H, Shen R, Zheng H, Yang G, Zhu Z; Chongqing Endocrine Hypertension Collaborative Team. Catheter-Based Adrenal Ablation Remits Primary Aldosteronism: A Randomized Medication-Controlled Trial. Circulation. 2021 Aug 17;144(7):580-582. doi: 10.1161/CIRCULATIONAHA.121.054318. Epub 2021 Aug 16. No abstract available. PMID 34398686
- [Result] Vaidya A, Carey RM. Evolution of the Primary Aldosteronism Syndrome: Updating the Approach. J Clin Endocrinol Metab. 2020 Dec 1;105(12):3771-83. doi: 10.1210/clinem/dgaa606. PMID 32865201
- [Result] Bouhanick B, Delchier MC, Lagarde S, Boulestreau R, Conil C, Gosse P, Rousseau H, Lepage B, Olivier P, Papadopoulos P, Trillaud H, Cremer A; for the ADERADHTA group. Radiofrequency ablation for adenoma in patients with primary aldosteronism and hypertension: ADERADHTA, a pilot study. J Hypertens. 2021 Apr 1;39(4):759-765. doi: 10.1097/HJH.0000000000002708. PMID 33196558
- [Result] Fowler AM, Burda JF, Kim SK. Adrenal artery embolization: anatomy, indications, and technical considerations. AJR Am J Roentgenol. 2013 Jul;201(1):190-201. doi: 10.2214/AJR.12.9507. PMID 23789675
- [Result] Williams TA, Lenders JWM, Mulatero P, Burrello J, Rottenkolber M, Adolf C, Satoh F, Amar L, Quinkler M, Deinum J, Beuschlein F, Kitamoto KK, Pham U, Morimoto R, Umakoshi H, Prejbisz A, Kocjan T, Naruse M, Stowasser M, Nishikawa T, Young WF Jr, Gomez-Sanchez CE, Funder JW, Reincke M; Primary Aldosteronism Surgery Outcome (PASO) investigators. Outcomes after adrenalectomy for unilateral primary aldosteronism: an international consensus on outcome measures and analysis of remission rates in an international cohort. Lancet Diabetes Endocrinol. 2017 Sep;5(9):689-699. doi: 10.1016/S2213-8587(17)30135-3. Epub 2017 May 30. PMID 28576687
- [Result] Kometani M, Yoneda T, Demura M, Karashima S, Mori S, Oe M, Sawamura T, Okuda R, Yamagishi M, Takeda Y. The Long-term Effect of Adrenal Arterial Embolization for Unilateral Primary Aldosteronism on Cardiorenovascular Protection, Blood Pressure, and the Endocrinological Profile. Intern Med. 2016;55(7):769-73. doi: 10.2169/internalmedicine.55.5196. Epub 2016 Apr 1. PMID 27041162
- [Result] Dong H, Zou Y, He J, Deng Y, Chen Y, Song L, Xu B, Gao R, Jiang X. Superselective adrenal arterial embolization for idiopathic hyperaldosteronism: 12-month results from a proof-of-principle trial. Catheter Cardiovasc Interv. 2021 May 1;97 Suppl 2:976-981. doi: 10.1002/ccd.29554. Epub 2021 Feb 19. PMID 33605538
- [Result] Hokotate H, Inoue H, Baba Y, Tsuchimochi S, Nakajo M. Aldosteronomas: experience with superselective adrenal arterial embolization in 33 cases. Radiology. 2003 May;227(2):401-6. doi: 10.1148/radiol.2272011798. Epub 2003 Apr 3. PMID 12676966
- [Result] Zhou Y, Wang D, Jiang L, Ran F, Chen S, Zhou P, Wang P. Diagnostic accuracy of adrenal imaging for subtype diagnosis in primary aldosteronism: systematic review and meta-analysis. BMJ Open. 2020 Dec 31;10(12):e038489. doi: 10.1136/bmjopen-2020-038489. PMID 33384386
- [Derived] Zhou Y, Liu S, Ji G, Yang C, Zhang L, Luo T, Huang F, Chen Z, Hou J, Wang P. Safety and efficacy of alcohol-mediated bilateral adrenal artery embolization in patients with idiopathic hyperaldosteronism: a 6-month follow-up of a randomized controlled trial. J Hum Hypertens. 2025 Jul;39(7):489-499. doi: 10.1038/s41371-025-01032-6. Epub 2025 Jun 4. PMID 40468047